CLINICAL TRIAL: NCT01182467
Title: Pilot Study in the Use of Positron Emission Tomography-Computed Tomography (PET-CT)in the Management of Crohn's Disease
Brief Title: Use of PET-CT in the Management of Crohn's Disease
Status: Terminated | Type: Observational
Why Stopped: PI left the institution
Sponsor: Columbia University (Other)
Responsible Party: Sponsor
Other Study IDs: AAAE8300
Record Dates: First submitted 2010-08-12; First posted 2010-08-16 (Estimated); Last update posted 2015-04-10 (Estimated); Status verified 2015-04

CONDITIONS: Crohn's Disease
Keywords: Inflammatory bowel disease, PET scan, Crohn's disease
MeSH Terms: conditions — Crohn Disease; Inflammatory Bowel Diseases

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Crohn's disease: Patients will receieve Radiation: PET-CT scan
  Interventions: Radiation: PET-CT scan

INTERVENTIONS:
Radiation: PET-CT scan — PET-CT scan performed at baseline to determine SUV-max
  Other Names: Positron emission tomography-computed tomography

SUMMARY:
Crohn's disease (CD) is an autoimmune disorder which affects over 700,000 people in the U.S. The disease can vary in severity and multiple drug classes are available to the disease depending on disease severity and complications. Our purpose will be to study how PET-CT scans can be used to better manage Crohn's Disease.

DETAILED DESCRIPTION:
Crohn's disease (CD) is a gastrointestinal autoimmune disease thought to result from exposure to luminal antigen. This exposure then results in a robust Th1 mediated immune response which is not downregulated, resulting in intestinal tissue injury. Crohn's disease most commonly involves the distal small intestine, a site that can be difficult to visualize given its central location within the gastrointestinal tract.

A substantial proportion of patients do not respond to any of the standard therapies. Over 40% of patients do not respond to an initial anti-TNF (biologic) agent and approximately 10% per year lose their response to these drugs. There is no standard definition of what constitutes a patient who has primary biologic failure.

Disease activity is measured by indices such as the Crohn's Disease Activity Index (CDAI). The CDAI includes a combination of clinical criteria and lab values. However, the CDAI is limited by reliance on subjective criteria, limiting the score's use as a valid measure of studying response to medical therapy. Clinically, reliance on CDAI can result in inappropriate continuation of an ineffective therapy resulting in worsening of underlying disease, and increasing risk of adverse reactions.

Small studies have demonstrated that PET scans may accurately quantify disease activity in Crohn's. We propose to study CD patients with active flares to assess for a correlation between PET activity and CDAI. Additionally, we will determine whether PET signal intensity is predictive of clinical response to therapy with biologic agents.

The study proposes to test the hypothesis that PET can be used to determine which CD patients with small bowel disease will be true responders (or nonresponders) to biologic therapy at week 12. The use of PET to determine response to biologic therapy in small bowel Crohn's disease would be novel.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Crohn's disease
* CDAI1>220
* Identification of small bowel disease based on an imaging study (CT scan, Abdominal ultrasound, MRI), colonoscopy, or histopathology 4. Need for initiation of biologic therapy to control disease process.

Exclusion Criteria:

* Abdominal surgery within 8 wks of study entry
* Change in dose of steroids or immunomodulators within 2wks of study entry
* Pregnancy
* Active bacterial infection or undrained abscess
* Any contraindications to initiation of AntiTNF therapy (i.e. latent tuberculosis).

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All adults between ages of 21-65 who have previously been diagnosed with Crohn's disease
Sampling Method: Non-Probability Sample
Enrollment: 5 (Actual)
Dates: Start 2011-02; Primary Completion 2013-09 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
Pravelence of PET activity with high CDAI score. | Baseline
  To determine whether baseline PET SUV-max correlates with response to biologic therapy, as measure by CDAI.

CONTACTS AND LOCATIONS:
Overall Officials: Arun Swaminath, MD, Principal Investigator — Columbia University; Masanori Ichise, MD, Principal Investigator — Columbia University
Locations (1):
- Columbia University Medical Center, New York, New York, United States